CLINICAL TRIAL: NCT07041515
Title: A Randomized, Multicenter Clinical Trial to Evaluate the Feasibility and Utility of a Postoperative Management App for Patients Undergoing Rectal Resection
Brief Title: Knowledge-enhanced Digital Intervention to Prevent Low Anterior Resection Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Dae Kyung Sohn, Principal Investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NCC2025-0022
Record Dates: First submitted 2025-04-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-04

CONDITIONS: Rectal Neoplasm
Keywords: rectal neoplasm; low anterior resection syndrome; Patient Reported Outcome
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- comparator (Active Comparator): Subjects classified as control group will receive educational materials.
  Interventions: Other: standard
- mobile app (Experimental): Subjects in the experimental group and pilot phase will install the management program app on their mobile phones and use it directly for 6 months.
  Interventions: Other: Mobile app

INTERVENTIONS:
Other: Mobile app — This study will be conducted in two stages, recruiting patients scheduled for low anterior resection and those scheduled for ostomy restoration after low anterior resection. The pilot stage study will recruit 20 subjects without randomization to evaluate the feasibility of the management program app, and the second stage study will be a parallel experimental-control study, recruiting approximately 300 research participants, 150 from each group.
  Patients scheduled for ostomy repair after low anterior resection and low anterior resection are required to fill out a consent form the day before, and participants are randomly assigned to one of two groups in a 1:1 ratio: the experimental group and the control group. Both groups are randomly assigned to four surveys. The types are three quality of life assessment questionnaires (QOL (EORTC QLQ-C30, CR-29, EQ-5D-L)) and a questionnaire related to bowel symptoms (LARS). However, patients undergoing ostomy repair are excluded from the preoperati
  Arms: mobile app
Other: standard — Subjects classified as control group will receive educational materials. One month and three months after surgery, a questionnaire related to bowel symptoms (LARS) will be administered by phone. The researcher will call the subjects and administer it according to the period. The results of the questionnaire related to bowel symptoms (LARS) administered by phone will be confirmed by the medical staff during outpatient treatment.
  Arms: comparator

SUMMARY:
Low anterior resection syndrome refers to changes in bowel habits such as frequent defecation, urgent defecation, and fecal incontinence, which result in decreased bowel function. It occurs very commonly after surgery for colorectal cancer, especially rectal cancer, and symptoms appear severely immediately after surgery, followed by a recovery process. It is known that symptoms improve significantly after one year of surgery, but in some patients, symptoms persist, which significantly affects the quality of life and causes social problems.

There is no established treatment method for low anterior resection syndrome, and accurate evaluation and customized treatment are required according to the patient's surgical or radiotherapy treatment content and symptoms. It is also important to monitor the change in symptoms during the treatment process, and a customized step-by-step treatment strategy for such patients is required. However, such a customized step-by-step treatment strategy for such patients is very complex, and there are no clear guidelines to date, and the research design for some clinical trials has been recently reported.

The purpose of this study was to develop an app-based Patient-Reported Outcome (PRO) standardized questionnaire for patients after rectal cancer surgery to systematically collect and monitor symptom information, establish a multidisciplinary management plan tailored to patients, and provide education and treatment to improve the quality of life of rectal cancer survivors. A management program utilizing a research device (app) can reduce the incidence of Major LARS after rectal cancer surgery compared to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20-70 years
2. Patients scheduled for anal-sparing rectal resection or stomy repair diagnosed with rectal cancer (within 15 cm from Anal Verge)
3. Patients with an expected survival period of 1 year or more
4. Patients or their primary caregivers use smartphones (apps)
5. Patients who are aware of their own status and can provide consent for this study

Exclusion Criteria:

1. If you are receiving chemotherapy or radiotherapy at the time of consent
2. If you are scheduled for major colectomy such as total colectomy or partial colectomy in addition to rectal resection
3. If you cannot be contacted by phone
4. If you cannot read and understand Korean
5. If you cannot provide consent based on clear and sufficient information

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2032-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of low anterior resection syndrome | 1 year after surgery
  The incidence of high-risk low anterior resection syndrome with a score of 30 to 42 in the bowel symptom questionnaire

SECONDARY OUTCOMES:
Symptom change | At patient registration and at 1, 3, 6, 12, 24, 36, and 60 months after surgery
  daily bowel frequency

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryoo SB, Ahn HM, Nam BH, Song YM, Sohn DK. K-LARS trial: protocol for a multicentre randomised controlled trial evaluating a knowledge-enhanced digital intervention to prevent low anterior resection syndrome in Korea. BMJ Open. 2025 Nov 29;15(11):e107819. doi: 10.1136/bmjopen-2025-107819. PMID 41320216